CLINICAL TRIAL: NCT04278365
Title: Affective Modulation of Positivity for Alcohol Use Disorder (AMP-A): Feasibility and Pilot Study
Brief Title: Affective Modulation of Positivity for Alcohol Use Disorder
Acronym: AMP-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-010
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-03

CONDITIONS: Anxiety; Depression; Alcohol Use Disorder
Keywords: Psychological
MeSH Terms: conditions — Anxiety Disorders; Depression; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMP-A (Experimental): Participants will complete 11, 90-minute sessions of positive affect training. The positive affect training will be conducted in an individual setting. Positive affect training directly targets reward and positive valence processing and has been shown by previous research to enhance positive affect (and decrease negative affect).
  Interventions: Behavioral: Positive affect training

INTERVENTIONS:
Behavioral: Positive affect training — Behavioral training involving position emotion enhancement
  Other Names: Affective Modulation of Positivity (AMP)

SUMMARY:
The proposed study is a pilot study examining the feasibility and potential utility of administering a psychosocial intervention termed Affective Modulation of Positivity (AMP) for individuals suffering from co-morbid depression or anxiety disorders and alcohol use disorder (AMP-A). The aims of this study are to (1) determine the feasibility and potential utility of administering AMP-A with individuals suffering from alcohol use disorders, (2) explore the potential impact of training on positive and negative affect, symptom severity, and functional disability, and (3) explore the potential impact of training on neural reactivity to reward and alcohol cues during functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
This study is a non-randomized, single-arm, single-site clinical trial conducted at Laureate Institute for Brain Research (LIBR) in Tulsa, OK. The primary objective for this study is to examine the feasibility and acceptability of conducting positive affect training with individuals suffering from substance use disorder. Primary outcome will include treatment completion rate; secondary outcome will include the score on a participant feedback questionnaire. The investigators hypothesize that the majority of participants (>60%) will complete all 11 sessions of the intervention and that participant feedback concerning the intervention will be at least moderately favorable on average.The secondary objective(s) is to explore the potential impact of training on positive and negative affect, symptom severity, and functional disability. The investigators hypothesize that positive affect will significantly increase from baseline to post-intervention, while negative affect, alcohol-related craving, and functional disability will significantly decrease. A tertiary objective is to explore the potential impact of training on behavioral and neural responses involving the processing of positively valenced or alcohol-related cues. The investigators hypothesize that activation with striatal and orbitofrontal cortex (OFC) regions to alcohol-UNrelated reward cues will increase from baseline to post-intervention, while striatal and OFC response to alcohol-related cues will decrease from baseline to post-intervention.

Participants will be asked to complete interview and pencil-and-paper questionnaires related to clinical symptoms, traits and personality characteristics, daily life function, and medical and mental health history at both pre- and post-intervention. Participants will also be asked to complete brief follow-up survey sessions 3 months after completing treatment. If there are participants who are only able to complete part of the intervention (i.e., only able to attend a few of the sessions) either due to their own wish to terminate or due to exclusion criteria or clinical concerns, they will only be asked to complete survey sessions for weeks that they attend. Neuroimaging procedures will be conducted at both pre- and post-intervention. Each neuroimaging session will last approximately 1.5-2.5 hours and will involve completion of self-report measures regarding current affective state and sleepiness and a functional MRI session during which participants will complete tasks related to reward processing and alcohol cue reactivity.

Following completion of baseline assessments, participants will be asked to complete 11 sessions of the positive affect intervention, conducted once or twice weekly and with each session lasting 1 - 1.5 hours. If the content of sessions is too much to cover for any one client, the intervention may be extended to 13 sessions as needed. Participants will be expected to complete all intervention sessions within 16 weeks of starting the first session. Each session will be completed as individual therapy sessions (i.e., one-on-one with a therapist). The positive affect intervention will involving positive emotion enhancement exercises established in prior studies, including noticing and amplifying positive emotions, practicing gratitude, engaging in acts of kindness, and pleasurable or meaningful activities, identifying strengths and values, being optimistic, engaging in activities meant to make others happy, and living life to its fullest. The investigators will use the protocol developed by Taylor et al. with modifications to specifically address alcohol use, based on previous work. The general structure of each session will follow standard cognitive behavioral treatment regimens as follows: (1) meet with clinician to review completion of the prior week's exercises, including self-monitoring forms of emotions and exercise completion; (2) identify and troubleshoot any issues that arose during exercise completion; (3) introduce material about a new positive emotion enhancement activity; (4) identify concrete exercises to implement for the upcoming week.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age between 18 and 55 years old.
2. Meeting diagnostic criteria for alcohol use disorder 41 according to the DSM-5.
3. Significant depression or anxiety symptoms as indexed by scoring Patient Health Questionnaire (PHQ-9) ≥ 10 and/or Overall Anxiety Severity and Impairment Scale (OASIS) ≥ 8.
4. Able to provide written informed consent.
5. Have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.
6. Completion of at least an 8th grade education, to help facilitate ability to engage in the written materials included in the Positive Affect Training.

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unwillingness or inability to complete any of the major aspects of the study protocol, including self-report or behavioral assessment. However, failing to complete some individual aspects of these assessment sessions will be acceptable (i.e., being unwilling to answer individual items on some questionnaires or being unwilling to complete a behavioral task).
2. Non-correctable vision or hearing problems.
3. No telephone or easy access to telephone.
4. Diagnosis of Schizophrenia spectrum, other psychotic disorders, or bipolar I disorder.
5. Active suicidal ideation with plan and intent to attempt suicide within the next month.
6. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
7. A positive test for drugs of abuse, including alcohol (breath test), cocaine, marijuana, opiates, amphetamines, methamphetamines, phencyclidine, benzodiazepines, barbiturates, methadone, and oxycodone at the time of baseline assessments. Participants will be asked to refrain from using alcohol within 24 hours prior to assessment sessions and to refrain from using marijuana within 48 hours of assessment sessions.
8. Current use of a medication or change in the dose or prescription of a medication within the 6 weeks prior to enrolling in the study that could potentially affect brain functioning (e.g., stimulants, anxiolytics, antipsychotics, mood stabilizers, anti-hypertensives). The current use of antidepressants (i.e., SSRIs) will not be excluded as long as the dose has remained consistent for 6 weeks prior to baseline assessment sessions. While individuals reporting use of benzodiazepines will be excluded; individuals with sporadic use (i.e., less than once per week) may be included, but will be asked to refrain from using within 72 hours prior to assessment sessions. Inclusion of individuals reporting other types of medications or supplements not listed or considered this far will be at the discretion of the PI according to evidence in the literature of it affecting brain function or brain blood flow.
9. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, and excessive caffeine intake > 1000 mg/day).
10. Concurrent engagement in psychosocial treatments that specifically target alcohol use disorder or mood/anxiety symptoms and began within 12 weeks of baseline assessments. Individuals concurrently receiving psychosocial treatments for other symptoms, or that are not specifically targeting symptoms (e.g., ongoing support groups) will not be excluded as long as the dose of treatment (i.e., frequency of sessions) has not changed significantly within 6 weeks prior to enrolling in the study.
11. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.
12. Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits, neurological disorders, or severe or unstable medical conditions that might be compromised by participation in the study (to be determined by primary care provider).
13. Severity of alcohol use disorder requiring more intensive treatment (i.e., intensive outpatient or residential), as determined by baseline assessments conducted by licensed clinicians.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Adherence and Acceptability Scale (AAS) | Post-intervention (within approximately 2 weeks after completing intervention)
  This measure assesses the acceptability and tolerability of the intervention. Scores may range from 10 to 70, with higher scores indicating greater acceptability of treatment and greater anticipated ability to adhere to it.
Distress/Endorsement Validation Scale (DEVS) | Post-intervention (within approximately 2 weeks after completing intervention)
  This measure assesses two factors, distress (7 items) and endorsement (3 items). The distress subscale score ranges from 7 to 63, with higher scores indicating more distress experienced during the intervention. The endorsement subscale ranges from 3 to 27, with higher scores indicating greater endorsement of the intervention.
Completion rate | Post-intervention (within approximately 2 weeks after completing intervention)
  Completion rate assessed as whether or not the participant completes all 11 sessions of intervention

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect and Well-being Scale | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses positive or rewarding affective experiences over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater positive affect and well-being.
Change in Alcohol Craving Questionnaire | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses four dimensions of alcohol craving. A total score ranges from 1-12, with higher scores indicating higher levels of alcohol craving.
Change in Positive and Negative Affect Schedule (PANAS) | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses factors related to positive and negative affect. Each of these factor scores range rom 10 to 50, with higher score indicates greater levels of positive and negative affect, respectively.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses symptoms of anxiety over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater symptoms of anxiety.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Scale | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses symptoms of depression over the past 7 days. The score is presented as a T score with a mean of 50 and standard deviation of 10, with higher scores indicating greater symptoms of depression.
Change in Sheehan Disability Scale | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measures assesses level of functional disability. Total score ranges from 0-30, with higher scores indicating greater impairment.
Change in alcohol use | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  As measured by self-reported drinks per day
Change in Snaith-Hamilton Please Scale (SHAPS) | Primary Endpoint: Post-treatment (i.e., within two weeks of completing the intervention). Secondary Endpoints: Three month follow-up (i.e., 12-15 weeks after completing the intervention)
  This measure assesses the ability to experience pleasure. Total scores range from 0 to 14, with a higher score indicating higher levels of anhedonia.

OTHER OUTCOMES:
Change in striatal responses during reward processing | Post-intervention (within approximately 2 weeks after completing intervention)
  Reward processing as measured by MID task
Change in striatal responses during alcohol cue processing | Post-intervention (within approximately 2 weeks after completing intervention)
  Alcohol cue processing as measured by alcohol cue task

CONTACTS AND LOCATIONS:
Overall Officials: Robin Aupperle, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taylor CT, Lyubomirsky S, Stein MB. Upregulating the positive affect system in anxiety and depression: Outcomes of a positive activity intervention. Depress Anxiety. 2017 Mar;34(3):267-280. doi: 10.1002/da.22593. Epub 2017 Jan 6. PMID 28060463
- [Derived] Akeman E, White E, Wolitzky-Taylor K, Santiago J, McDermott TJ, DeVille DC, Stewart JL, Paulus M, Taylor CT, Aupperle RL. Amplification of Positivity Therapy for Co-occurring Alcohol Use Disorder with Depression and Anxiety Symptoms: Pilot Feasibility Study and Case Series. Behav Modif. 2022 Sep;46(5):1021-1046. doi: 10.1177/01454455211030506. Epub 2021 Jul 12. PMID 34253077